CLINICAL TRIAL: NCT03830957
Title: Randomized Clinical Trial of Ivabradine to Reduce Heart Rate Prior to Coronary CT-angiography in Advanced Heart Failure: Comparison With β-Blocker
Brief Title: Efficacy and Safety of Ivabradine to Reduce Heart Rate Prior to Coronary CT-angiography in Advanced Heart Failure: Comparison With β-Blocker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HFRC_01
Record Dates: First submitted 2018-11-26; First posted 2019-02-05 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; CT Angiography; Ischemic Cardiomyopathy; Non-ischemic Cardiomyopathy; Heart Failure, Systolic; Heart Failure，Congestive; Heart Failure, Diastolic; Heart Rate Low
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic; Bradycardia | interventions — Ivabradine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Active Comparator)
  Interventions: Drug: Ivabradine
- metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Ivabradine — 7.5 mg oral single dose if the heart rate would not reach to 60/minute then give another dose, 7.5 mg
  Arms: Ivabradine
Drug: Metoprolol — 5 mg oral single dose if the heart rate would not reach to 60/minute then give another dose, 5 mg
  Arms: metoprolol

SUMMARY:
The aim of this study is to compare the effects of Ivabradine and metoprolol to reduce heart rate prior to coronary CT angiography in patients with advanced heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Sinus rhythm
* Heart rate >60/min

Exclusion Criteria:

* Atrial fibrillation
* Any contraindication for beta-blocker use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 30 minutes before and after coronary CT angiography
  Changing heart rate during imaging study

SECONDARY OUTCOMES:
Dyspnea | 30 minutes before and after coronary CT angiography and 6 months later
  Shortness of breath, or "dyspnea", is the most famous symptom of left ventricular failure. It typically appears during strenuous activities, and progresses to ordinary activities, less than ordinary activities and ultimately resting state. The severity is categorized as above (FC 1 to 4)
Functional calss | 30 minutes before and after coronary CT angiography and 6 months later
  Heart Failure severity has been classified according to New York Heart Association (NYHA) to:
  * Class I: No limitation of physical activity. Ordinary physical activity does not cause symptoms of HF.
  * Class II: Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in symptoms of HF.
  * Class III: Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes symptoms of HF.
  * Class IV: Unable to perform any physical activity without symptoms of HF, or symptoms of HF at rest.
Blood pressure, systolic and diastolic | 30 minutes before and after coronary CT angiography and 6 months later
  The amount of blood pressure measured by sphygmomanometer
Sleep quality | Before CT angiography and 6 months later
  The rate of disturbed sleep measured as better than before, Worse than before, and No change
  There are no standard classification for severity of this symptom. In our study, we measure this symptom as :
  * Better than before (1)
  * Worse than before (2)
  * No change (0)
Appetite | Before CT angiography and 6 months later
  The rate of changing in appetite level measured as better than before, Worse than before, and No change
  Loss of appetite is a common symptom of heart failure. There are no standard classification for severity of this symptom. In our study, we measure this symptom as :
  * Better than before (1)
  * Worse than before (2)
  * No change (0)
Prolonged bradycardia | 30 minutes before and after coronary CT angiography
  Persistence of Bradycardia more than 6 hours is called prolonged bradycardia.
Hypotension | 30 minutes before and after coronary CT angiography
  Systolic less than 80 mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Amin, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided